CLINICAL TRIAL: NCT00734539
Title: Fluconazole Prophylaxis for the Prevention of Candidiasis in Infants < 750 Grams Birth
Brief Title: Fluconazole Prophylaxis for the Prevention of Candidiasis in Infants Less Than 750 Grams Birthweight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daniel Benjamin (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Thrasher Research Fund (Other); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Daniel Benjamin, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00001538; 1R01HD057956-01 (NIH); Pro00017720 (Other: DUMC)
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Candidiasis
Keywords: Candida; Neonate; Fluconazole; Prophylaxis; Colonization; Resistance
MeSH Terms: conditions — Candidiasis; Torulopsis | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): fluconazole 6mg/kg IV or PO twice weekly for 6 weeks
  Interventions: Drug: fluconazole
- 2 (Placebo Comparator): Placebo IV or PO twice weekly for 6 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fluconazole — 6mg/kg IV/PO twice weekly for a total of up to 12-13 doses
  Other Names: Diflucan
  Arms: 1
Drug: placebo — normal saline (IV) or 3 parts Ora Plus oral suspension vehicle and 1 part simethicone suspension (PO): will be given twice weekly PO/IV for a total of up to 12-13 doses
  Arms: 2

SUMMARY:
The most common etiology of infection-related death or neurodevelopmental impairment in neonates with birthweight <750 g is invasive candidiasis. Over 70% of the premature neonates who develop invasive candidiasis will die or suffer severe, permanent neurologic impairment. Fluconazole has been commonly used off-label in the neonatal intensive care unit, but definitive recommendations for its use in the nursery have been hampered by the limited number of well-designed trials. In neonates weighing <750 g, appropriate dosing is not known, definitive safety and long-term follow up trials have not been completed, and there have not been well-powered trials conducted to establish the efficacy of the product using mortality as part of the primary endpoint. Three recent proof-of-concept studies suggest that fluconazole will be safe and effective, and a recently completed pharmacokinetic study is providing data to give preliminary dosing guidance. The next logical step in drug development is proposed by this research: to conduct a pivotal trial to determine the safety and efficacy of fluconazole in premature neonates with 2-year neurodevelopmental follow-up assessment.

362 neonates, with a birthweight <750g, were randomized at 33 US centers, to twice weekly fluconazole (6 mg/kg) or placebo for the first 6 weeks of life. The primary efficacy endpoint will be Candida-free survival at study day 49. The research will establish definitive dosing, safety, and efficacy of fluconazole; it will also provide critical information on the effects of fluconazole on neurodevelopmental impairment and antifungal resistance.

Potential Impact:

Approximately 17,000 neonates are born <750 grams each year in the United States. Over 5000 will die or develop invasive Candida infections. Demonstrating safety and efficacy of fluconazole in preterm neonates will improve the survivability and long term outcomes for these neonates.

DETAILED DESCRIPTION:
362 subjects were randomized to the study at 33 US sites. Final study visits of Month 18-22 corrected age long term follow up were completed. Study database is locked.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from the legally authorized representative.
* > 48 hours of age and < 120 hours old at time of first drug administration
* < 750 g birth weight
* Negative blood cultures for Candida

Exclusion Criteria:

* History of a hypersensitivity or severe vasomotor reaction to any azole
* receiving antifungal therapy for suspected/proven invasive fungal infection
* medical condition, in the opinion of the Investigator, may create an unacceptable additional risk
* diagnosed with invasive candidiasis or congenital Candida infection.
* liver failure (AST and ALT > 250 U/L)
* renal failure (creatinine > 2 mg/dL)
* major lethal congenital or genetic anomalies
* triplet or higher multiple gestations

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel K Benjamin, MD MPH PhD, Principal Investigator — Duke Univerisity Medical Center, Duke Clinical Research Institute
Locations (33):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - University of California-San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Shands Jacksonville Medical Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Riley Hospital, Indianapolis, Indiana
  - Memorial Hospital, South Bend, Indiana
  - Wesley Medical Center, Wichita, Kansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Wayne State University, Detroit, Michigan
  - University of Minnesota, Fairview Medical Center, Minneapolis, Minnesota
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - West Jersey Hospital - Voorhees, Voorhees Township, New Jersey
  - Brookdale University Medical Center, Brooklyn, New York
  - Kings County Hospital Center, Brooklyn, New York
  - SUNY Dowstate Medical Center, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Oregon Health Sciences Center, Portland, Oregon
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Cooks Children's Medical Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - University of Texas - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In December 2018, after receiving IRB's approval, the team submitted the de-identified study dataset and redacted study documents to the NICHD Data and Specimen Hub (DASH).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: DASH was published in December 2018. DASH is managed by NICHD for future research.
Access Criteria: DASH is managed by NICHD.
URL: https://dash.nichd.nih.gov/Study/19811

REFERENCES:
- [Derived] Benjamin DK Jr, Hudak ML, Duara S, Randolph DA, Bidegain M, Mundakel GT, Natarajan G, Burchfield DJ, White RD, Shattuck KE, Neu N, Bendel CM, Kim MR, Finer NN, Stewart DL, Arrieta AC, Wade KC, Kaufman DA, Manzoni P, Prather KO, Testoni D, Berezny KY, Smith PB; Fluconazole Prophylaxis Study Team. Effect of fluconazole prophylaxis on candidiasis and mortality in premature infants: a randomized clinical trial. JAMA. 2014 May 7;311(17):1742-9. doi: 10.1001/jama.2014.2624. PMID 24794367
- [Derived] Moran C, Smith PB, Cohen-Wolkowiez M, Benjamin DK Jr. Clinical trial design in neonatal pharmacology: effect of center differences, with lessons from the Pediatric Oncology Cooperative Research experience. Clin Pharmacol Ther. 2009 Dec;86(6):589-91. doi: 10.1038/clpt.2009.175. PMID 19915602

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluconazole: fluconazole 6mg/kg IV or PO twice weekly for 6 weeks
  fluconazole: 6 mg/kg PO/IV twice weekly x 14 doses
- Placebo: Placebo IV or PO twice weekly for 6 weeks
  placebo: placebo: normal saline (IV) or 3 parts Ora Plus oral suspension vehicle and 1 part simethicone suspension (PO): will be given twice weekly PO/IV for 14 doses
Period: Main Study
Arm/Group | Fluconazole | Placebo
Started | 189 | 173
Completed | 152 (Number of subjects who participated through hospital discharge or study end) | 138 (Number of subjects who participated through hospital discharge or study end)
Not Completed | 37 | 35
Not completed — Death | 33 | 32
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Enrolled in error; ineligible | 1 | 0
Period: Long Term Follow up
Arm/Group | Fluconazole | Placebo
Started | 152 | 138
Completed | 118 (Number of participants who completed the 18-22 months follow-up) | 107 (Number of participants who completed the 18-22 months follow-up)
Not Completed | 34 | 31

BASELINE CHARACTERISTICS:
Population: Infants who received at least 1 dose of study drug (Modified Intent-to-Treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluconazole | Placebo | Total
Number analyzed (Participants) | 188 | 173 | 361
Age, Continuous [Median (Inter-Quartile Range); unit: days] — Postnatal age at randomization
  days | 3 [3 to 4] | 3 [2 to 4] | 3 [2 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 98 | 207
  Male | 79 | 75 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 25 | 46
  Not Hispanic or Latino | 167 | 148 | 315
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — 2 participants specified a race as "other" which is not pre-specified in this list of races.
  Participants
    American Indian or Alaska Native | 10 | 7 | 17
    Asian | 3 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 102 | 94 | 196
    White | 73 | 70 | 143
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 2 | 2
birth weight [Median (Inter-Quartile Range); unit: grams] | 653 [570 to 700] | 640 [573 to 700] | 650 [570 to 700]
Gestational Age at Birth [Median (Inter-Quartile Range); unit: weeks] | 25 [24 to 26] | 25 [24 to 26] | 25 [24 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Death or Candidiasis
Description: The primary endpoint for the study is death or candidiasis.
  1. Death prior to study day 49.
  2. Candidiasis prior to study day 49
     1. Definite: isolation of Candida from normally sterile body fluid (blood, CSF, urine [obtained via sterile catheterization or suprapubic tap], peritoneal fluid).
     2. Probable:
     i. > 5 days of consecutive antifungal therapy
     AND both:
     ii. Thrombocytopenia <150,000/mm3 iii. Positive Candida culture from nonsterile site (ETS, bag urine)
Time Frame: study day 49
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 31 | 37

2. Secondary Outcome: Neurodevelopmental Impairment
Description: Bayley-III cognition composite score of less than 70, blindness, deafness, or cerebral palsy
Time Frame: 18-22 months corrected gestational age
Population: Attended the follow-up visit and had complete data on composite endpoint
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 87 | 84
participants | 27 | 23

3. Secondary Outcome: Candidiasis
Description: Definite or probable
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 8 | 19

4. Secondary Outcome: Stage II or Higher Necrotizing Enterocolitis
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 25 | 23

5. Secondary Outcome: Focal Intestinal Perforation
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 16 | 9

6. Secondary Outcome: Chronic Lung Disease
Time Frame: 36 weeks corrected gestational age
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 114 | 93

7. Secondary Outcome: Patent Ductus Arterious Requiring Surgical Ligation
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 46 | 43

8. Secondary Outcome: Periventricular Leukomalacia
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 10 | 6

9. Secondary Outcome: Retinopathy of Prematurity Requiring Laser Surgery
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 29 | 25

10. Secondary Outcome: Length of Hospitalization
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
days | 113 [90 to 148] | 107 [88 to 128]

11. Secondary Outcome: Positive Bacterial Infection From a Sterile Site
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Fluconazole: fluconazole 6mg/kg IV or PO twice weekly for 6 weeks
  fluconazole: 6mg/kg IV/PO twice weekly for a total of up to 12-13 doses
- Placebo: Placebo IV or PO twice weekly for 6 weeks
  placebo: normal saline (IV) or 3 parts Ora Plus oral suspension vehicle and 1 part simethicone suspension (PO): will be given twice weekly for a total of up to 12-13 doses
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 109 | 100

12. Secondary Outcome: Intraventricular Hemorrhage
Description: Grade 3 or 4
Time Frame: prior to hospital discharge, up to 15 ½ months
Population: Modified intent-to-treat; only subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo IV or PO twice weekly for 6 weeks
  placebo: normal saline (IV) or 3 parts Ora Plus oral suspension vehicle and 1 part simethicone suspension (PO): will be given twice weekly PO/IV for a total of up to 12-13 doses
Arm/Group | Fluconazole | Placebo
Number analyzed (Participants) | 188 | 173
participants | 33 | 31

ADVERSE EVENTS:
Time Frame: From time of first dose of study drug until 30 days following the last dose, up to approximately 10 weeks
Arm/Group | Fluconazole | Placebo
Serious Adverse Events (participants affected / at risk) | 83/188 | 68/173
Other Adverse Events (participants affected / at risk) | 1/188 | 1/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluconazole (N=188) | Placebo (N=173)
Necrotising Enterocolitis Neonatal (Gastrointestinal disorders) | 27 | 28
Intestinal Perforation (Gastrointestinal disorders) | 12 | 6
Meconium Ileus (Gastrointestinal disorders) | 2 | 0
Colonic Stenosis (Gastrointestinal disorders) | 1 | 0
Ileal Perforation (Gastrointestinal disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Peritoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal Prolapse (Gastrointestinal disorders) | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Sepsis Neonatal (Infections and infestations) | 5 | 12
Staphylococcal Sepsis (Infections and infestations) | 4 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Arthritis Bacterial (Infections and infestations) | 1 | 0
Candida Sepsis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Group B Streptococcus Neonatal Sepsis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Neonatal Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Neonatal Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Neonatal Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Intraventricular Haemorrhage Neonatal (Nervous system disorders) | 2 | 3
Hydrocephalus (Nervous system disorders) | 2 | 1
Convulsion Neonatal (Nervous system disorders) | 1 | 1
Cerebral Ventricle Dilatation (Nervous system disorders) | 1 | 0
Bradycardia Neonatal (Cardiac disorders) | 2 | 1
Neonatal Cardiac Failure (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest Neonatal (Cardiac disorders) | 0 | 1
Neonatal Hypotension (Vascular disorders) | 1 | 3
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Vena Cava Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Neonatal Multi-Organ Failure (General disorders) | 1 | 3
Infusion Site Extravasation (General disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 1
Renal Failure Neonatal (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 1 | 1
Ileal Atresia (Congenital, familial and genetic disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Adrenal Insufficiency (Endocrine disorders) | 2 | 0
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 1
Bilirubin Conjugated Increased (Investigations) | 1 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0
Retinopathy of Prematurity (Eye disorders) | 0 | 1
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluconazole (N=188) | Placebo (N=173)
Hyperbilirubinaemia Neonatal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes